CLINICAL TRIAL: NCT01059565
Title: Phase 3b Randomized, Double-Blind, Placebo-Controlled Two-Part Trial to Assess the Safety and Efficacy of Continuous Aztreonam for Inhalation Solution (AZLI) in Subjects With Cystic Fibrosis (CF) and Chronic Burkholderia Species Infection
Brief Title: Safety and Efficacy Study of Aztreonam for Inhalation Solution (AZLI) in Patients With Cystic Fibrosis and Chronic Burkholderia Species Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-205-0127
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Cystic Fibrosis; Burkholderia Infections
Keywords: Cystic Fibrosis; Aztreonam Lysine; lung infection; Burkholderia; CFQ-R; inhaled antibiotic
MeSH Terms: conditions — Cystic Fibrosis; Burkholderia Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZLI (Experimental): Participants were randomized to receive AZLI for up to 24 weeks and may have continued to receive AZLI during the open-label phase for up to an additional 24 weeks.
  Interventions: Drug: AZLI
- Placebo (Placebo Comparator): Participants were randomized to receive placebo to match AZLI for up to 24 weeks and may have switched to AZLI during the open-label phase for up to 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZLI — Aztreonam for inhalation solution (AZLI; 75 mg aztreonam/52.5 mg lysine monohydrate) was administered three times a day, with at least 4 hours between doses, using the investigational nebulizer.
  Arms: AZLI
Drug: Placebo — Placebo to match AZLI (lactose and sodium chloride) was administered three times a day, with at least 4 hours between doses, using the investigational nebulizer.
  Arms: Placebo

SUMMARY:
The purpose of this research study was to determine if an experimental drug called Aztreonam for Inhalation Solution (AZLI) was safe and effective to treat Burkholderia lung infections in patients with cystic fibrosis (CF).

Spirometry was used to assess pulmonary function, and the revised Cystic Fibrosis Questionnaire (CFQ-R) was used to assess quality of life. The CFQ-R is a validated, patient-reported outcome tool used to measure health-related quality of life for children and adults with CF.

The study consisted of a 24-week randomized phase, and a 24-week open-label phase. Primary and secondary efficacy analyses were conducted for the 24-week randomized phase only. Safety data were collected for both the randomized and open-label phases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 6 years of age
2. Subjects with CF as diagnosed by one of the following:

   * Documented sweat chloride ≥ 60 milliequivalent (mEq)/L by quantitative pilocarpine iontophoresis test
   * Documented sweat sodium ≥ 60 mmol/L
   * Two well-characterized genetic mutations in the CF transmembrane conductance regulator (CFTR) gene
   * Abnormal nasal potential difference (NPD) with accompanying symptoms characteristic of CF
3. Chronic infection with Burkholderia spp. defined by:

   * One sputum (or bronchoalveolar lavage) culture positive for Burkholderia spp. within 6 months prior to baseline assessment,
   * At least 50% of sputum (or bronchoalveolar lavage) cultures collected at least one month apart over the previous 12 months prior to baseline assessment positive for Burkholderia spp. (minimum of 2 positive cultures), and
   * At least one positive sputum (or bronchoalveolar lavage) culture (obtained at any point in time) confirmed to be Burkholderia spp. by the Cystic Fibrosis Foundation (CFF) Burkholderia cepacia Research Laboratory and Repository at the University of Michigan (or equivalent Canadian reference laboratory).
4. Concomitant aerosolized antibiotic treatment: subjects receiving intermittent (alternating month on/month off) aerosolized antibiotic treatment were eligible, but must have been at least 1 week into their off-treatment cycle at the time of baseline assessment. Subjects receiving continuous aerosolized antibiotic treatment were eligible without restriction on their aerosolized antibiotic treatment.
5. Chest radiograph, computed tomography (CT), or magnetic resonance imaging (MRI) (most recent, obtained within 90 days of screening) without significant acute findings (eg, infiltrates [lobar or diffuse interstitial], pleural effusion, pneumothorax), and no significant intercurrent illness; chronic, stable findings (eg, chronic scarring or atelectasis) were allowed.
6. Subjects (and parent/guardian as required) must have been able to provide written informed consent/assent prior to any study-related procedures,
7. Ability to perform reproducible pulmonary function tests
8. Sexually active females of childbearing potential must have agreed to use a highly effective method of contraception during heterosexual intercourse throughout the study period and for 30 days following discontinuation of study drug. A highly effective method of birth control was defined as a method that would result in a low failure rate (ie, less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), or a vasectomized partner.

Exclusion Criteria:

1. Administration of any investigational drug or use of any investigational device within 28 days of randomization/baseline and within six half-lives of the investigational drug (whichever is longer)
2. Administration of AZLI treatment within the 28 days prior to randomization/baseline
3. Known local or systemic hypersensitivity to monobactam antibiotics
4. History of lung transplantation
5. Abnormal renal or hepatic function results at most recent test within the previous 90 days, defined as:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of the normal range (ULN)
   * Serum creatinine > 2 times ULN
6. Known portal hypertension or complications of CF hepatopathy
7. Positive urine pregnancy test (confirmed by serum pregnancy test) at screening; all women of childbearing potential were tested
8. Any female of childbearing potential who was lactating or not practicing a highly effective method of birth control as defined in the protocol
9. Any serious or active medical or psychiatric illness which, in the opinion of the investigator, would have interfered with subject treatment, assessment or compliance with the protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, MD, Study Director — Gilead Sciences
Locations (35):
- United States (34):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Denver, Colorado
  - Hartford, Connecticut
  - Wilmington, Delaware
  - Jacksonville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Glenview, Illinois
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - New Hyde Park, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Richmond, Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 34 sites in the United States and 1 site in Canada. The first participant was screened on 22 February 2010. The last participant observation was on 28 December 2010.
Pre-assignment Details: 102 participants were screened and 101 were randomized. Of those participants randomized, 100 received at least one dose of study drug, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- AZLI: Aztreonam for inhalation solution (AZLI; 75 mg aztreonam/52.5 mg lysine monohydrate) was administered three times a day, with at least 4 hours between doses, using the investigational nebulizer. After the 24-week randomized phase, participants continued to receive AZLI during the open-label phase.
- Placebo: Placebo to match AZLI (lactose and sodium chloride) was administered three times a day, with at least 4 hours between doses, using the investigational nebulizer. After the 24-week randomized phase, participants switched to AZLI during the open-label phase.
Period: 24-Week Randomized Phase
Arm/Group | AZLI | Placebo
Started | 49 | 52
Randomized and Treated | 48 | 52
Completed | 39 | 45
Not Completed | 10 | 7
Not completed — Randomized but not treated | 1 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Noncompliance with Study Drug Regimen | 1 | 5
Period: 24-Week Open-Label Phase
Arm/Group | AZLI | Placebo
Started | 39 | 45
Completed | 34 | 42
Not Completed | 5 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Worsening health (physician decision) | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Subject noncompliance | 1 | 0
Not completed — Unable to clean device (hospitalization) | 0 | 1
Not completed — Pulmonologist/participant decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants were randomized and received at least one dose of study drug.
Groups:
- AZLI: Aztreonam for inhalation solution (AZLI; 75 mg aztreonam/52.5 mg lysine monohydrate) was administered three times a day, with at least 4 hours between doses, for up 48 weeks using the investigational nebulizer.
- Placebo: Placebo to match AZLI (lactose and sodium chloride) was administered three times a day, with at least 4 hours between doses, for up 48 weeks using the investigational nebulizer.
- Total: Total of all reporting groups
Arm/Group | AZLI | Placebo | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (10.3) | 24.7 (10.0) | 26.3 (10.2)
Age, Customized [Number; unit: participants]
  ≥ 6 to ≤ 12 years | 3 | 3 | 6
  > 12 to < 18 years | 3 | 8 | 11
  ≥ 18 years | 42 | 41 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 26 | 35 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 48 | 51 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African Heritage | 1 | 2 | 3
  White | 46 | 50 | 96
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 45 | 49 | 94
  Canada | 3 | 3 | 6
Forced expiratory volume in 1 second (FEV1) percent predicted [Mean (Standard Deviation); unit: percentage of FEV1 % predicted] — FEV1 % predicted is defined as FEV1 % of the patient divided by the average FEV1 % in the population for any person of similar age, sex and body composition.
  percentage of FEV1 % predicted | 60.67 (21.71) | 52.59 (23.71) | 56.47 (23.02)
FEV1 [Mean (Standard Deviation); unit: liters] — FEV1 is defined as the maximal volume of air that can be exhaled in 1 second.
  liters | 2.13 (0.93) | 1.93 (0.96) | 2.02 (0.95)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: liters] — FVC is defined as the volume of air that can forcibly be blown out after taking a full breath.
  liters | 3.23 (1.18) | 2.99 (1.14) | 3.11 (1.16)
Forced expiratory flow 25% to 75% (FEF25-75) [Mean (Standard Deviation); unit: liters per second] — FEF25-75 is defined as the forced expiratory flow from 25% to 75% of the FVC.
  liters per second | 1.33 (0.95) | 1.31 (1.22) | 1.32 (1.09)
Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) Score [Mean (Standard Deviation); unit: units on a scale] — Respiratory symptoms (e.g., coughing, congestion, wheezing) were assessed with the CFQ-R Respiratory Symptoms Scale (RSS). The range of scores (units) is 0 to 100 with higher scores indicating fewer symptoms.
  units on a scale | 58.3 (21.4) | 59.0 (17.6) | 58.6 (19.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 21.9 (4.5) | 20.7 (3.2) | 21.3 (3.9)
Burkholderia spp colony-forming units (CFU) in sputum [Mean (Standard Deviation); unit: log_10 CFU per gram] — Participants in the Full Analysis Set with evaluable assessments for Burkholderia spp. CFU in sputum at baseline were analyzed, which included 30 in the AZLI group, 32 in the placebo group, and 62 total.
  log_10 CFU per gram | 6.39 (2.47) | 6.41 (2.52) | 6.40 (2.48)

OUTCOME MEASURES:

1. Primary Outcome: AUCave of Relative Change in FEV1 % Predicted From Baseline to Week 24
Description: The relative change (AUCave) in FEV1 % predicted from baseline to Week 24 was analyzed. FEV1 % predicted is defined as FEV1 % of the patient divided by the average FEV1 % in the population for any person of similar age, sex and body composition. AUCave is the calculated area under the curve corrected for baseline and adjusted by the number of days on study through Week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change in FEV1% predicted
Groups:
- AZLI: AZLI was administered three times a day, with at least 4 hours between doses, for up 48 weeks using the investigational nebulizer.
- Placebo: Placebo to match AZLI was administered three times a day, with at least 4 hours between doses, for up 48 weeks using the investigational nebulizer.
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 48 | 52
percent change in FEV1% predicted | 0.16 (1.50) | -0.75 (1.43)
Statistical Analysis 1: Comparison: AZLI vs Placebo; The primary analysis was a test for superiority. Null hypothesis was no difference between the AZLI and placebo treatment groups versus the alternative hypothesis that there was a difference. A sample size of 50 participants per group provided at least 80% power to detect an 8.5% difference in mean AUCave of relative change from baseline in FEV1 % predicted through Week 24 using a two-sided 0.05-level test, assuming a common standard deviation of 15; Test type: Superiority or Other; p = 0.663, ANCOVA — To correct for multiplicity, a family alpha spending rule was used to control the type 1 error rate of alpha=0.05. A gate-keeping procedure to control family-wise Type 1 error was established a priori for primary and key secondary endpoints; Baseline was included as a covariate in this model; Difference in least squares mean (LSM) = 0.91, 95% CI 2-sided [-3.24 to 5.06]

2. Secondary Outcome: Total Number of Systemic and/or Inhaled Antibiotic Courses for Respiratory Events
Description: The total number of systemic and/or inhaled antibiotic courses for respiratory events from baseline to Week 24 was analyzed. A single antibiotic course may represent the use of multiple antibiotics.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Number; unit: antibiotic treatment courses
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 48 | 52
antibiotic treatment courses | 54 | 73
Statistical Analysis 1: Comparison: AZLI vs Placebo; The primary analysis was a test for superiority. Null hypothesis was no difference between the AZLI and placebo treatment groups versus the alternative hypothesis that there was a difference; Test type: Superiority or Other; p = 0.4158, Negative binomial regression — To correct for multiplicity, a family alpha spending rule was used to control the type 1 error rate of alpha=0.05; The negative binomial regression model included an offset parameter which accounted for potential differing study durations due to discontinuations

3. Secondary Outcome: AUCave of Change in CFQ-R RSS Scores From Baseline to Week 24
Description: The change (AUCave) in CFQ-R RSS scores from baseline to Week 24 was analyzed.
  The range of scores (units) within the RSS domain is 0 to 100 with higher scores indicating fewer symptoms.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 45 | 52
units on a scale | 2.97 (1.70) | 2.79 (1.58)
Statistical Analysis 1: Comparison: AZLI vs Placebo; Null hypothesis was that there was no difference between the AZLI and placebo treatment groups versus the alternative hypothesis that there was a difference; Test type: Superiority or Other; p = 0.939, ANCOVA — To correct for multiplicity, a family alpha spending rule was used to control the type 1 error rate of alpha=0.05; The AUCs of changes from baseline were compared between treatment groups using ANCOVA methods with baseline value as a covariate; Difference in LSM = 0.18, 95% CI 2-sided [-4.43 to 1.78]

4. Secondary Outcome: AUCave of Relative Change From Baseline to Week 24 in FEV1
Description: The relative change (AUCave) from baseline to Week 24 in mean (SE) FEV1 was analyzed. FEV1 is defined as the maximal volume of air that can be exhaled in 1 second.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in FEV1 (liters)
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 47 | 52
percent change in FEV1 (liters) | 0.36 (1.49) | -0.41 (1.42)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.711, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in LSM = 0.77, 95% CI 2-sided [-3.33 to 4.86]

5. Secondary Outcome: AUCave of Relative Change From Baseline to Week 24 in FVC
Description: The relative change (AUCave) from baseline to Week 24 in mean (SE) FVC was analyzed. FVC is defined as the volume of air that can forcibly be blown out after taking a full breath.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in FVC (liters)
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 47 | 52
percent change in FVC (liters) | 0.77 (1.42) | 0.17 (1.35)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.762, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in LSM = 0.60, 95% CI 2-sided [-3.30 to 4.49]

6. Secondary Outcome: AUCave of Relative Change From Baseline to Week 24 in FEF25-75
Description: The relative change (AUCave) from baseline to Week 24 in mean (SE) FEF25-75 was analyzed. FEF25-75 is defined as the forced expiratory flow from 25% to 75% of the FVC.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in FEF25-75 (liters/sec)
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 47 | 52
percent change in FEF25-75 (liters/sec) | 1.40 (2.37) | -0.55 (2.25)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.553, ANCOVA; [statistical method as in outcome 3, analysis 1]; Difference in LSM = 1.95, 95% CI 2-sided [-4.54 to 8.44]

7. Secondary Outcome: AUCave of the Change From Baseline to Week 24 in Physical Functioning Score as Assessed by the CFQ-R
Description: The change (AUCave) from baseline to Week 24 in the physical functioning score as assessed by the CFQ-R was analyzed.
  The range of scores (units) in the CFQ-R physical functioning domain is 0 to 100 with higher scores indicating better QOL.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 46 | 52
units on a scale | 1.06 (1.57) | -1.93 (1.48)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.170, ANCOVA; Baseline was included as a covariate in this model; Difference in LSM = 2.99, 95% CI 2-sided [-1.20 to 7.28]

8. Secondary Outcome: AUCave of the Change From Baseline to Week 24 in Weight Score as Assessed by the CFQ-R
Description: The change (AUCave) from baseline to Week 24 in the weight score as assessed by the CFQ-R was analyzed.
  The range of scores (units) in the CFQ-R weight domain is 0 to 100 with higher scores indicating better QOL.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 44 | 47
units on a scale | 0.54 (2.90) | 3.11 (2.80)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.528, ANCOVA; Baseline was included as a covariate in this model; Difference in LSM = -2.57, 95% CI 2-sided [-10.62 to 5.49]

9. Secondary Outcome: AUCave of the Change From Baseline to Week 24 in Treatment Burden Score as Assessed by the CFQ-R
Description: The change (AUCave) from baseline to Week 24 in the treatment burden score as assessed by the CFQ-R was analyzed.
  The range of scores (units) in the CFQ-R treatment burden domain is 0 to 100 with higher scores indicating better QOL.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 46 | 52
units on a scale | -2.73 (1.73) | -6.35 (1.62)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.132, ANCOVA; Baseline was included as a covariate in this model; Difference in LSM = 3.62, 95% CI 2-sided [-1.11 to 8.34]

10. Secondary Outcome: Change in BMI From Baseline to Week 24
Description: The change in BMI from baseline to Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 39 | 45
kg/m^2 | 0.34 (0.16) | 0.21 (0.15)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.531, Mixed Models Analysis; P-value was based on a Mixed-Effect Model Repeated Measure model that included terms for treatment, visit, baseline, and treatment/visit interaction; Difference in LSM = 0.14, 95% CI 2-sided [-0.29 to 0.56]

11. Secondary Outcome: Change in Burkholderia Spp. CFU in Sputum From Baseline to Week 24
Description: The change in Burkholderia spp. CFU in sputum from baseline to Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available change data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: log_10 CFU per gram of sputum
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 15 | 20
log_10 CFU per gram of sputum | 1.41 (0.58) | 0.48 (0.50)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.232, ANCOVA; Baseline was included as a covariate in this model; Difference in LSM = 0.93, 95% CI 2-sided [-0.62 to 2.48]

12. Secondary Outcome: Percentage of Days Participants Used Antibiotics
Description: The percentage of days participants used antibiotics from baseline to Week 24 was analyzed. Antibiotics ongoing at baseline or started on or after first dose date were included in the analysis. A single antibiotic course could represent the use of multiple antibiotics. Days of antibiotic use included unique days.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 47 | 52
percentage of days | 44.4 (35.2) | 56.3 (34.8)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.103, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Percent of Days Hospitalized
Description: The percentage of days hospitalized from baseline to Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 48 | 52
percentage of days | 4.9 (10.3) | 4.8 (8.7)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.646, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Percentage of Missed School or Work Days
Description: The percentage of days participants missed school or work from baseline to Week 24 was analyzed.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 32 | 40
percentage of days | 1.9 (3.3) | 4.7 (7.2)
Statistical Analysis 1: Comparison: AZLI vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.284, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline to Week 24
Groups:
- AZLI: For the reporting of Adverse Events, this group includes participants who were randomized to receive AZLI at baseline, and were analyzed from Baseline to Week 24.
- Placebo: For the reporting of Adverse Events, this group includes participants who were randomized to receive placebo at baseline, and were analyzed from Baseline to Week 24.
- AZLI/AZLI: For the reporting of Adverse Events, this group includes participants who were randomized to receive AZLI at baseline and continued to receive an up to an additional 24 weeks of AZLI treatment during the open-label phase, and were analyzed from Week 24 to Week 48.
- Placebo/AZLI: For the reporting of Adverse Events, this group includes participants who were randomized to receive placebo at baseline and switched AZLI for up to 24 weeks of treatment during the open-label phase, and were analyzed from Week 24 to Week 48.
Arm/Group | AZLI | Placebo | AZLI/AZLI | Placebo/AZLI
Serious Adverse Events (participants affected / at risk) | 17/48 | 21/52 | 19/39 | 24/45
Other Adverse Events (participants affected / at risk) | 46/48 | 46/52 | 39/39 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=48) | Placebo (N=52) | AZLI/AZLI (N=39) | Placebo/AZLI (N=45)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Infective pulmonary exacerbation of cycstic fibrosis (Infections and infestations) | 10 | 6 | 8 | 11
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 7 | 14 | 9 | 9
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholethiasis (General disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Haematspermia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (N=48) | Placebo (N=52) | AZLI/AZLI (N=39) | Placebo/AZLI (N=45)
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 3
Chest discomfort (General disorders) | 13 | 8 | 6 | 9
Chest pain (General disorders) | 7 | 1 | 13 | 10
Chills (General disorders) | 6 | 2 | 8 | 3
Constipation (Gastrointestinal disorders) | 3 | 3 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 32 | 31 | 34
Decreased appetite (Metabolism and nutrition disorders) | 8 | 6 | 8 | 7
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 4 | 6
Dizziness (Nervous system disorders) | 5 | 3 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 17 | 21
Exercise tolerance decreased (General disorders) | 5 | 1 | 1 | 3
Fatigue (General disorders) | 10 | 11 | 14 | 12
Forced expiratory volume decreased (Investigations) | 2 | 3 | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 | 17 | 11 | 8
Headache (Nervous system disorders) | 6 | 7 | 8 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1
Insomnia (Psychiatric disorders) | 4 | 1 | 4 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 16 | 14
Nausea (Gastrointestinal disorders) | 11 | 10 | 7 | 7
Non-cardiac chest pain (General disorders) | 3 | 3 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 15 | 15
Pain (General disorders) | 6 | 2 | 3 | 5
Paranasal sinus hypersectretion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 3
Pulmonary function test decreased (Investigations) | 5 | 8 | 3 | 9
Pyrexia (General disorders) | 19 | 17 | 16 | 19
Rales (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 7 | 6
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 14 | 13 | 11
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0
Rhinorrheoa (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 10 | 9
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 12 | 3
Sinus headache (Nervous system disorders) | 8 | 3 | 9 | 1
Sinusitis (Infections and infestations) | 1 | 4 | 4 | 5
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 23 | 20 | 19 | 14
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 2 | 2
Vomiting (Gastrointestinal disorders) | 7 | 5 | 4 | 4
Weight decreased (Investigations) | 3 | 3 | 4 | 7
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 8 | 6
Asthenia (General disorders) | 4 | 3 | 2 | 4
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 2 | 3
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Breath sounds abmormal (Investigations) | 0 | 0 | 4 | 2
Vitamin D decreased (Investigations) | 0 | 0 | 4 | 2
Oxygen saturation decreased (Investigations) | 0 | 0 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 3
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 5
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years